CLINICAL TRIAL: NCT00064038
Title: Phase III Trial Comparing Dexamethasone (DEX) to the Combination of DEX + CC-5013 in Patients With Previously Untreated Multiple Myeloma
Brief Title: S0232 Dexamethasone With or Without Lenalidomide in Treating Patients With Previously Untreated Stage I, Stage II, or Stage III Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S0232; U10CA032102 (NIH); S0232 (Other: SWOG)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Results first posted 2013-07-17 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Myeloma; Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Dexamethasone; Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive induction therapy comprising oral dexamethasone (DM) on days 1-4, 9-12, and 17-20 and oral lenalidomide on days 1-28. Treatment repeats every 35 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance therapy comprising oral DM on days 1-4 and 15-18 and oral lenalidomide on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dexamethasone; Drug: lenalidomide
- Arm II (Active Comparator): Patients receive induction therapy comprising DM as in arm I induction and oral placebo on days 1-28. Treatment repeats as in arm I induction. Some patients may then receive maintenance therapy comprising oral DM as in arm I maintenance and oral placebo on days 1-21. Courses repeat as in arm I maintenance.
  Interventions: Drug: dexamethasone; Other: placebo

INTERVENTIONS:
Drug: dexamethasone — Given orally
Drug: lenalidomide — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as dexamethasone use different ways to stop cancer cells from dividing so they stop growing or die. Lenalidomide may stop the growth of multiple myeloma by stopping blood flow to the tumor. It is not yet known whether dexamethasone is more effective with or without lenalidomide in treating multiple myeloma.

PURPOSE: This randomized phase III trial is studying dexamethasone and lenalidomide to see how well they work compared to dexamethasone alone in treating patients with previously untreated stage I, stage II, or stage III multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the progression-free survival of patients with previously untreated stage I, II, or III multiple myeloma treated with dexamethasone with or without lenalidomide.
* Compare the overall response rate in patients treated with these regimens.
* Compare the major response rate (indicated by greater than 75% decrease in M-protein) in patients treated with these regimens.
* Compare the overall survival and time to best response in patients treated with these regimens.
* Compare the toxicity profile of these regimens, including thrombotic complications, in these patients.
* Compare the effect of these regimens on gene expression and proteomic analysis in these patients.

OUTLINE: This is a randomized, double-blind, crossover, multicenter study. Patients are stratified according to disease stage by the International Staging System (I vs II vs III) and Zubrod performance status (0-1 vs 2-3). Patients are randomized to 1 of 2 treatment arms.

Arm I

* Induction therapy: Patients receive oral dexamethasone (DM) on days 1-4, 9-12, and 17-20 and oral lenalidomide on days 1-28. Treatment repeats every 35 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
* Maintenance therapy: Patients receive oral DM on days 1-4 and 15-18 and oral lenalidomide on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Arm II

* Induction therapy: Patients receive DM as in arm I induction and oral placebo on days 1-28. Treatment repeats as in arm I induction.

Patients with responding or stable disease proceed to maintenance therapy. Patients with disease progression during induction therapy cross over and receive unblinded treatment with DM and lenalidomide as in arm I induction. Patients with responding or stable disease after unblinded induction therapy receive unblinded maintenance therapy with DM and lenalidomide as in arm I maintenance.

* Maintenance therapy: Patients receive oral DM as in arm I maintenance and oral placebo on days 1-21. Courses repeat as in arm I maintenance.

Patients with disease progression during maintenance therapy cross over and receive unblinded treatment with DM and lenalidomide as in arm I induction. Patients with responding or stable disease after unblinded induction therapy proceed to unblinded maintenance therapy with DM and lenalidomide as in arm I maintenance.

Patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 500 patients (250 per treatment arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Previously untreated multiple myeloma

  * Stage I, II, or III disease by the International Staging System
* Measurable M-protein as defined by 1 of the following:

  * Serum M-protein at least 1.0 g/dL by serum protein electrophoresis or immunoelectrophoresis
  * Urinary M-protein excretion at least 200 mg/24 hours
* No nonsecretory multiple myeloma
* Not planning to undergo future autologous stem cell transplantation

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-3* NOTE: *Zubrod 3 allowed only if multiple myeloma is the central cause of disability

Life expectancy

* Not specified

Hematopoietic

* Platelet count at least 80,000/mm^3*
* Absolute neutrophil count at least 1,000/mm^3*
* Hemoglobin at least 9 g/dL* (epoetin alfa or transfusion allowed) NOTE: *Unless due to greater than 50% marrow involvement by myeloma on biopsy

Hepatic

* AST/ALT no greater than 3 times upper limit of normal* NOTE: *Values outside of this range are allowed at the investigator's discretion

Renal

* Creatinine no greater than 2.5 mg/dL* NOTE: *Values outside of this range are allowed at the investigator's discretion

Cardiovascular

* No New York Heart Association class III or IV heart failure
* No myocardial infarction within the past 6 months
* No poorly controlled hypertension

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 4 weeks before, during, and for 4 weeks after study treatment

  * Female patients must use 2 reliable forms of contraception simultaneously
  * Male patients must use effective barrier contraception
* No uncontrolled active infection requiring IV antibiotics
* No poorly controlled diabetes mellitus that would preclude ability to take oral glucocorticoids
* No other serious medical condition that would preclude study participation
* No psychiatric illness that would preclude study participation
* No other malignancy within the past 3 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Must be able to take aspirin by mouth at a dose of 325 mg per day or enoxaparin subcutaneously at a dose of 40 mg per day as a form of thrombotic prophylaxis, except if already on therapeutic anticoagulant medication

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior interferon or thalidomide

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Prior high-dose dexamethasone allowed provided duration of administration was no more than 4 days

Radiotherapy

* Prior localized radiotherapy allowed provided it was not to the sole site of evaluable disease

Surgery

* Not specified

Other

* No prior treatment for clinically significant ventricular cardiac arrhythmias
* Concurrent bisphosphonates allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2004-11; Primary Completion 2008-10 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Zonder, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah

REFERENCES:
- [Result] Zonder JA, Crowley JJ, Bolejack V, et al.: A randomized Southwest Oncology Group study comparing dexamethasone (D) to lenalidomide + dexamethasone (LD) as treatment of newly-diagnosed multiple myeloma (NDMM): impact of cytogenetic abnormalities on efficacy of LD, and updated overall study results. [Abstract] J Clin Oncol 26 (Suppl 15): A-8521, 2008.
- [Result] Zonder JA, Crowley J, Hussein MA, et al.: Superiority of lenalidomide (Len) plus high-dose dexamethasone (HD) compared to HD alone as treatment of newly-diagnosed multiple myeloma (NDMM): results of the randomized, double-blinded, placebo-controlled SWOG trial S0232. [Abstract] Blood 110 (11): A-77, 2007.
- [Derived] Zonder JA, Crowley J, Hussein MA, Bolejack V, Moore DF Sr, Whittenberger BF, Abidi MH, Durie BG, Barlogie B. Lenalidomide and high-dose dexamethasone compared with dexamethasone as initial therapy for multiple myeloma: a randomized Southwest Oncology Group trial (S0232). Blood. 2010 Dec 23;116(26):5838-41. doi: 10.1182/blood-2010-08-303487. Epub 2010 Sep 27. PMID 20876454

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 15, 2004 and April 2, 2007, 198 patients were enrolled at 41 cooperative medical institutions.
Groups:
- Lenalidomide+Dexamethasone: Patients receive induction therapy comprising oral dexamethasone (DM) on days 1-4, 9-12, and 17-20 and oral lenalidomide on days 1-28. Treatment repeats every 35 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance therapy comprising oral DM on days 1-4 and 15-18 and oral lenalidomide on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Dexamethasone: Patients receive induction therapy comprising DM as in arm I induction and oral placebo on days 1-28. Treatment repeats as in arm I induction. Some patients may then receive maintenance therapy comprising oral DM as in arm I maintenance and oral placebo on days 1-21. Courses repeat as in arm I maintenance.
- Crossover to Lenalidomide+Dexamethasone: Patients who have progressive or relapsed disease or who experience unacceptable toxicity attributable to dexamethasone dosing level -2 while on blinded treatment, will be unblinded. Patients shown to have been randomized to DEX + Placebo will proceed with crossover registration and Open-Label Induction with DEX + CC-5013or with open-label CC-5013 alone if they are unblinded due to dexamethasone toxicity.
  Patients receive induction therapy comprising oral dexamethasone (DM) on days 1-4, 9-12, and 17-20 and oral lenalidomide on days 1-28. Treatment repeats every 35 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance therapy comprising oral DM on days 1-4 and 15-18 and oral lenalidomide on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Initial Randomization
Arm/Group | Lenalidomide+Dexamethasone | Dexamethasone | Crossover to Lenalidomide+Dexamethasone
Started | 100 | 98 | 0
Eligible and Analyzable | 97 | 95 | 0
Safety Population | 96 | 94 | 0
Completed | 0 (The study was closed early per recommedation of the Data Safety Monitoring Committee.) | 0 (The study was closed early per recommedation of the Data Safety Monitoring Committee.) | 0
Not Completed | 100 | 98 | 0
Period: Crossover to Lenalidomide+Dexamethasone
Arm/Group | Lenalidomide+Dexamethasone | Dexamethasone | Crossover to Lenalidomide+Dexamethasone
Started | 0 | 0 (See Crossover to Lenalidomide+Dexamethasone Arm.) | 42
Eligible and Analyzable | 0 | 0 (See Crossover to Lenalidomide+Dexamethasone Arm.) | 40
Safety Population | 0 | 0 (See Crossover to Lenalidomide+Dexamethasone Arm.) | 40
Completed | 0 | 0 (See Crossover to Lenalidomide+Dexamethasone Arm.) | 40
Not Completed | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide+Dexamethasone | Dexamethasone | Total
Number analyzed (Participants) | 97 | 95 | 192
Age, Continuous [Median (Full Range); unit: years]
  Overall | 64.9 [36.9 to 89.0] | 63.1 [37.6 to 87.0] | 64.6 [36.9 to 89.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 40 | 84
  Male | 53 | 55 | 108

OUTCOME MEASURES:

1. Secondary Outcome: Toxicity
Description: Compare the toxicity profile of these regimens, including thrombotic complications, in these patients, based on CTCAE v. 3.0.
Time Frame: From time of initiating study treatment until discontinuation of study treatment or of open-label REVLIMID + LOW DOSE DEX, whichever comes last, up to 5 years
Population: All participants receiving at least one dose of induction therapy
Measure: Number; unit: Participants
Groups:
- Lenalidomide and Dexamethasone; Crossover to Rev+Dex: Patients receive induction therapy comprising oral dexamethasone (DM) on days 1-4, 9-12, and 17-20 and oral lenalidomide on days 1-28. Treatment repeats every 35 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients then receive maintenance therapy comprising oral DM on days 1-4 and 15-18 and oral lenalidomide on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Lenalidomide and Dexamethasone | Dexamethasone | Crossover to Rev+Dex
Number analyzed (Participants) | 96 | 94 | 40
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 1 | 1 | 0
  AST, SGOT | 2 | 0 | 0
  Albumin, serum-low (hypoalbuminemia) | 1 | 0 | 2
  Anorexia | 2 | 1 | 1
  Apnea | 1 | 0 | 0
  Arthritis (non-septic) | 1 | 0 | 0
  Aspiration | 1 | 0 | 0
  Ataxia (incoordination) | 0 | 1 | 0
  Bilirubin (hyperbilirubinemia) | 0 | 0 | 1
  CNS cerebrovascular ischemia | 1 | 2 | 2
  Calcium, serum-high (hypercalcemia) | 0 | 1 | 0
  Calcium, serum-low (hypocalcemia) | 7 | 2 | 3
  Cardiopulmonary arrest, cause unknown (non-fatal) | 1 | 0 | 0
  Cataract | 1 | 1 | 2
  Cognitive disturbance | 1 | 1 | 0
  Colitis | 0 | 0 | 1
  Colitis, infectious (e.g., Clostridium difficile) | 0 | 0 | 1
  Confusion | 1 | 0 | 0
  Constipation | 0 | 2 | 1
  Creatinine | 0 | 0 | 1
  Cystitis | 0 | 1 | 0
  Dehydration | 1 | 0 | 3
  Dermatology/Skin-Other (Specify) | 0 | 1 | 0
  Diarrhea | 5 | 1 | 1
  Dizziness | 1 | 1 | 2
  Dyspnea (shortness of breath) | 4 | 2 | 0
  Edema: limb | 0 | 1 | 2
  Encephalopathy | 0 | 0 | 1
  Fatigue (asthenia, lethargy, malaise) | 19 | 12 | 8
  Febrile neutropenia | 1 | 0 | 1
  Fever in absence of neutropenia, ANC lt1.0x10e9/L | 1 | 1 | 0
  Fracture | 0 | 1 | 0
  Gastritis (including bile reflux gastritis) | 0 | 0 | 1
  Gastrointestinal-Other (Specify) | 1 | 0 | 0
  Glomerular filtration rate | 0 | 0 | 1
  Glucose, serum-high (hyperglycemia) | 5 | 18 | 2
  Glucose, serum-low (hypoglycemia) | 1 | 0 | 0
  Heartburn/dyspepsia | 0 | 1 | 0
  Hemoglobin | 6 | 5 | 6
  Hemorrhage, CNS | 1 | 0 | 0
  Hemorrhage, GI - Colon | 1 | 0 | 0
  Hypertension | 0 | 3 | 0
  Hypotension | 3 | 0 | 0
  Hypoxia | 4 | 1 | 1
  INR (of prothrombin time) | 1 | 2 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 1 | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Bronchus | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 5 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Up aerodigest | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Upper airway | 1 | 2 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Bladder | 2 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Bronchus | 0 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Colon | 1 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 1 | 3 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Skin | 2 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - UTI | 2 | 2 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Up airway | 3 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Wound | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils -Nerve-cran | 0 | 0 | 1
  Infection with unknown ANC - Lung (pneumonia) | 1 | 0 | 0
  Infection with unknown ANC - Upper airway NOS | 1 | 1 | 0
  Infection-Other (Specify) | 0 | 1 | 0
  Insomnia | 4 | 6 | 0
  Joint-function | 1 | 0 | 0
  Left ventricular diastolic dysfunction | 0 | 0 | 1
  Left ventricular systolic dysfunction | 1 | 0 | 0
  Leukocytes (total WBC) | 14 | 5 | 4
  Lymphopenia | 10 | 5 | 8
  Mood alteration - agitation | 1 | 1 | 1
  Mood alteration - anxiety | 1 | 1 | 0
  Mood alteration - depression | 11 | 8 | 2
  Mucositis/stomatitis (clinical exam) - Oral cavity | 0 | 1 | 0
  Muscle weakness, not d/t neuropathy - Extrem-lower | 1 | 3 | 1
  Muscle weakness, not d/t neuropathy - body/general | 9 | 4 | 3
  Musculoskeletal/Soft Tissue-Other (Specify) | 0 | 2 | 0
  Nausea | 2 | 1 | 0
  Neuropathy: motor | 0 | 1 | 0
  Neuropathy: sensory | 3 | 4 | 0
  Neutrophils/granulocytes (ANC/AGC) | 21 | 6 | 7
  Ocular/Visual-Other (Specify) | 1 | 0 | 1
  Ophthalmoplegia/diplopia (double vision) | 0 | 1 | 0
  Opportunistic inf associated w/gt=Gr 2 lymphopenia | 2 | 0 | 1
  PTT (Partial thromboplastin time) | 0 | 1 | 0
  Pain - Abdomen NOS | 0 | 2 | 0
  Pain - Back | 1 | 2 | 1
  Pain - Bladder | 0 | 0 | 1
  Pain - Bone | 1 | 3 | 0
  Pain - Extremity-limb | 1 | 0 | 0
  Pain - Head/headache | 0 | 1 | 0
  Pain - Joint | 3 | 1 | 0
  Pain - Muscle | 3 | 1 | 1
  Pain - Pain NOS | 1 | 0 | 0
  Pain - Stomach | 0 | 1 | 0
  Pain-Other (Specify) | 0 | 1 | 1
  Pancreatic endocrine: glucose intolerance | 0 | 1 | 0
  Perforation, GI - Colon | 1 | 0 | 0
  Perforation, GI - Small bowel NOS | 0 | 1 | 0
  Phosphate, serum-low (hypophosphatemia) | 5 | 4 | 2
  Platelets | 7 | 4 | 3
  Pneumonitis/pulmonary infiltrates | 3 | 2 | 2
  Potassium, serum-low (hypokalemia) | 6 | 2 | 3
  Prolonged QTc interval | 1 | 0 | 0
  Proteinuria | 1 | 0 | 0
  Pulmonary/Upper Respiratory-Other (Specify) | 1 | 0 | 0
  Rash/desquamation | 1 | 1 | 1
  Rash: acne/acneiform | 0 | 1 | 1
  Rash: erythema multiforme | 0 | 0 | 1
  Renal failure | 0 | 1 | 2
  SVT and nodal arrhythmia - Atrial fibrillation | 0 | 2 | 0
  Sodium, serum-high (hypernatremia) | 0 | 1 | 0
  Sodium, serum-low (hyponatremia) | 3 | 2 | 3
  Somnolence/depressed level of consciousness | 0 | 0 | 1
  Speech impairment (e.g., dysphasia or aphasia) | 0 | 0 | 1
  Syncope (fainting) | 1 | 0 | 0
  Thrombosis/embolism (vascular access-related) | 2 | 0 | 0
  Thrombosis/thrombus/embolism | 19 | 5 | 5
  Thrombotic microangiopathy | 1 | 0 | 0
  Thyroid function, low (hypothyroidism) | 1 | 0 | 0
  Tinnitus | 1 | 0 | 0
  Vision-blurred vision | 2 | 3 | 1
  Vomiting | 2 | 1 | 0
  Weight loss | 0 | 0 | 1

2. Primary Outcome: Progression-Free Survival
Description: Progression is defined as a > 25% increase from baseline in myeloma protein production or other signs of disease progression such as hypercalcemia, etc.
  In patients with a confirmed Partial Remission, Remission, or Complete Remission, relapse is defined as the first occurrence of any of the following: 1) a myeloma protein increase by than 100% from the lowest level recorded on study, provided the absolute magnitude of this increase is at least 1g/dL for a serum monoclonal protein or at least 500 mg/24 hrs of urine M-protein; 2) a myeloma protein increase above the response criteria for Partial Remission, with the same requirements for the absolute magnitude of the protein increase; 3)reappearance of any myeloma peak that had disappeared while on protocol treatment, provided it meets the same requirements listed above; 4) increase in the size and number of lytic bone lesions recognized on radiographs.
Time Frame: From date of initial registration to date of progression/relapse of disease or death from any cause, whichever came first, up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide+Dexamethasone | Dexamethasone
Number analyzed (Participants) | 97 | 95
percentage of participants | 78 [70 to 78] | 52 [41 to 62]

ADVERSE EVENTS:
Time Frame: Report through 1/13/2009 to match data reported in MS.
Arm/Group | Lenalidomide and Dexamethasone | Dexamethasone | Crossover to Rev+Dex
Serious Adverse Events (participants affected / at risk) | 41/96 | 21/94 | 14/40
Other Adverse Events (participants affected / at risk) | 91/96 | 90/94 | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide and Dexamethasone (N=96) | Dexamethasone (N=94) | Crossover to Rev+Dex (N=40)
Hemoglobin (Blood and lymphatic system disorders) | 3 | 2 | 1
Cardiac General-Other (Specify) (Cardiac disorders) | 1 | 0 | 0
Cardiac-ischemia/infarction (Cardiac disorders) | 2 | 0 | 0
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 3 | 0 | 0
Supraventricular (SVT) and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1 | 2 | 0
SVT and nodal arrhythmia - Atrial tachycardia/paroxysmal atrial tachycardia (PAT) (Cardiac disorders) | 0 | 0 | 1
Ocular/Visual-Other (Specify) (Eye disorders) | 0 | 0 | 1
Vision-blurred vision (Eye disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 | 0 | 0
Fistula, GI - Abdomen, not otherwise specified (NOS) (Gastrointestinal disorders) | 1 | 0 | 0
Fistula, GI - Colon/cecum/appendix (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhage, GI - Colon (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhage, GI - Lower GI NOS (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Obstruction, GI - Colon (Gastrointestinal disorders) | 0 | 0 | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 0 | 2 | 0
Perforation, GI - Colon (Gastrointestinal disorders) | 1 | 1 | 0
Stricture/stenosis (incl anastomotic), Esophagus (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Death not associated with CTCAE term - Death, not otherwise specified (NOS) (General disorders) | 1 | 1 | 0
Edema: limb (General disorders) | 0 | 1 | 0
Extremity-lower (gait/walking) (General disorders) | 0 | 1 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 | 2 | 0
Pain - Pain NOS (General disorders) | 1 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 1 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Bronchus (Infections and infestations) | 1 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 2 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Up aerodigest (Infections and infestations) | 1 | 0 | 0
Inf w/normal absolute neutrophil count (ANC) or Gr 1-2 neutrophils - Ab NOS (Infections and infestations) | 1 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Bladder (Infections and infestations) | 2 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Colon (Infections and infestations) | 1 | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 2 | 2 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 1 | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 2 | 2 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Up airway (Infections and infestations) | 1 | 0 | 0
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1 | 0 | 0
Infection-Other (Specify) (Infections and infestations) | 0 | 1 | 0
Opportunistic inf associated w/gt=Gr 2 lymphopenia (Infections and infestations) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 3 | 0
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 2 | 0 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 0 | 0 | 1
Cardiac troponin T (cTnT) (Investigations) | 1 | 0 | 0
Creatinine (Investigations) | 3 | 0 | 0
International normalized ratio (INR) (of prothrombin time) (Investigations) | 1 | 1 | 0
Leukocytes (total white blood cell count (WBC)) (Investigations) | 3 | 0 | 0
Lymphopenia (Investigations) | 2 | 1 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 3 | 0 | 0
Platelets (Investigations) | 2 | 0 | 1
Prolonged QTc interval (Investigations) | 1 | 0 | 0
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 0 | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 | 1 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 | 0 | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 | 0 | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 0 | 2
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Musculoskeletal/Soft Tissue-Other (Specify) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Death - Disease progression, not otherwise specified (NOS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Central nervous system (CNS) cerebrovascular ischemia (Nervous system disorders) | 1 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Ocular/Visual-Other (Specify) (Nervous system disorders) | 0 | 0 | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 | 0 | 1
Syncope (fainting) (Nervous system disorders) | 0 | 1 | 1
Mood alteration - depression (Psychiatric disorders) | 0 | 1 | 0
Cystitis (Renal and urinary disorders) | 0 | 1 | 0
Glomerular filtration rate (Renal and urinary disorders) | 0 | 0 | 1
Hemorrhage, GU - Urinary, not otherwise specified (NOS) (Renal and urinary disorders) | 0 | 1 | 0
Obstruction, GU - Ureter (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Hemorrhage, pulmo/upper resp- Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pain - Pleura (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1
Hematoma (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0
Phlebitis (including superficial thrombosis) (Vascular disorders) | 1 | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 13 | 4 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide and Dexamethasone (N=96) | Dexamethasone (N=94) | Crossover to Rev+Dex (N=40)
Hemoglobin (Blood and lymphatic system disorders) | 62 | 63 | 31
Palpitations (Cardiac disorders) | 0 | 5 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 5 | 0
Cataract (Eye disorders) | 6 | 0 | 3
Ocular/Visual-Other (Specify) (Eye disorders) | 0 | 0 | 2
Vision-blurred vision (Eye disorders) | 12 | 9 | 5
Constipation (Gastrointestinal disorders) | 43 | 34 | 19
Diarrhea (Gastrointestinal disorders) | 44 | 29 | 9
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 5 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 | 8 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 18 | 12 | 2
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 7 | 10 | 5
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 7 | 11 | 0
Nausea (Gastrointestinal disorders) | 36 | 24 | 11
Pain - Abdomen, not otherwise specified (NOS) (Gastrointestinal disorders) | 9 | 7 | 3
Pain - Dental/teeth/peridontal (Gastrointestinal disorders) | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 11 | 10 | 0
Edema: head and neck (General disorders) | 0 | 13 | 0
Edema: limb (General disorders) | 36 | 35 | 13
Fatigue (asthenia, lethargy, malaise) (General disorders) | 74 | 71 | 31
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 7 | 15 | 3
Pain - Chest/thorax NOS (General disorders) | 8 | 8 | 3
Pain-Other (Specify) (General disorders) | 5 | 0 | 3
Rigors/chills (General disorders) | 6 | 8 | 2
Inf (clin/microbio) w/Gr 3-4 neuts - Upper airway (Infections and infestations) | 0 | 5 | 0
Inf w/normal absolute neutrophil count (ANC) or Gr 1-2 neutrophils - Bronchus (Infections and infestations) | 0 | 0 | 3
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 5 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Sinus (Infections and infestations) | 0 | 0 | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 9 | 5 | 2
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 0 | 0 | 4
Inf w/normal ANC or Gr 1-2 neutrophils - Up airway (Infections and infestations) | 23 | 15 | 5
Infection with unknown ANC - Sinus (Infections and infestations) | 0 | 0 | 2
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 0 | 0 | 2
Infection with unknown ANC - Upper airway, not otherwise specified (NOS) (Infections and infestations) | 6 | 0 | 0
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 0 | 0 | 2
Bruising (in absence of Gr 3-4 thrombocytopenia) (Injury, poisoning and procedural complications) | 0 | 0 | 2
Alanine aminotransferase (ALT), serum glutamic pyruvic transaminase (SGPT) (Investigations) | 17 | 14 | 4
Aspartate aminotransferase (AST), serum glutamic oxaloacetic transaminase (SGOT) (Investigations) | 12 | 11 | 7
Alkaline phosphatase (Investigations) | 17 | 10 | 4
Bilirubin (hyperbilirubinemia) (Investigations) | 10 | 5 | 4
Creatinine (Investigations) | 22 | 20 | 12
Leukocytes (total WBC) (Investigations) | 51 | 28 | 20
Lymphopenia (Investigations) | 28 | 24 | 16
Metabolic/Laboratory-Other (Specify) (Investigations) | 0 | 6 | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 42 | 22 | 15
Platelets (Investigations) | 35 | 24 | 16
Weight gain (Investigations) | 7 | 8 | 4
Weight loss (Investigations) | 22 | 14 | 3
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 24 | 21 | 13
Anorexia (Metabolism and nutrition disorders) | 24 | 20 | 11
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 5 | 11 | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 43 | 38 | 19
Dehydration (Metabolism and nutrition disorders) | 10 | 12 | 7
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 53 | 59 | 22
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 9 | 0 | 3
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 12 | 9 | 2
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 14 | 9 | 5
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 | 10 | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 35 | 21 | 18
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 6 | 5 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 11 | 23 | 8
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 0 | 0 | 2
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 5 | 8 | 4
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 23 | 15 | 5
Musculoskeletal/Soft Tissue-Other (Specify) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 34 | 25 | 13
Pain - Bone (Musculoskeletal and connective tissue disorders) | 16 | 21 | 8
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 14 | 12 | 6
Pain - Joint (Musculoskeletal and connective tissue disorders) | 21 | 21 | 12
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 21 | 12 | 10
Pain - Neck (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 22 | 18 | 8
Memory impairment (Nervous system disorders) | 0 | 0 | 2
Neuropathy: motor (Nervous system disorders) | 5 | 8 | 4
Neuropathy: sensory (Nervous system disorders) | 49 | 32 | 9
Ocular/Visual-Other (Specify) (Nervous system disorders) | 0 | 0 | 2
Pain - Head/headache (Nervous system disorders) | 13 | 12 | 5
Taste alteration (dysgeusia) (Nervous system disorders) | 26 | 15 | 5
Tremor (Nervous system disorders) | 10 | 10 | 2
Confusion (Psychiatric disorders) | 7 | 8 | 2
Insomnia (Psychiatric disorders) | 34 | 49 | 8
Mood alteration - agitation (Psychiatric disorders) | 7 | 9 | 2
Mood alteration - anxiety (Psychiatric disorders) | 10 | 9 | 0
Mood alteration - depression (Psychiatric disorders) | 30 | 23 | 9
Incontinence, urinary (Renal and urinary disorders) | 0 | 0 | 2
Pain - Bladder (Renal and urinary disorders) | 0 | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 3
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 15 | 5
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 19 | 18 | 0
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 2
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 5 | 11 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 0 | 0
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 6 | 5 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 22 | 17 | 11
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 10 | 13 | 2
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Flushing (Vascular disorders) | 0 | 0 | 2
Hot flashes/flushes (Vascular disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 9 | 8 | 2
Hypotension (Vascular disorders) | 12 | 5 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 10 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No